CLINICAL TRIAL: NCT00962156
Title: Effects of Hydroxyethyl Starch 130/0.4 Compared With Balanced Crystalloid Solution on Mortality and Kidney Failure in Patients With Severe Sepsis
Brief Title: Scandinavian Starch for Severe Sepsis/Septic Shock Trial
Acronym: 6S
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anders Perner (Other)
Collaborators: Rigshospitalet, Denmark (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other); B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor-Investigator, Anders Perner, Chairman, Scandinavian Critical Care Trials Group
Organization: Scandinavian Critical Care Trials Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-262; EudraCT no. 2009-010104-28
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis; Shock; Fluid therapy; Plasma expanders
MeSH Terms: conditions — Sepsis; Shock, Septic; Shock | interventions — Hydroxyethyl Starch Derivatives; LHFPL6 protein, human; Ringerfundin; sterofundin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HES 130/0.4 (Experimental): Volume expansion
  Interventions: Drug: 6% Hydroxyethyl starch 130/0.4
- Ringer acetate (Active Comparator): Volume expansion
  Interventions: Drug: Ringers acetate

INTERVENTIONS:
Drug: 6% Hydroxyethyl starch 130/0.4 — Infusion for volume expansion in the ICU
  Other Names: 6% Tetraspan
  Arms: HES 130/0.4
Drug: Ringers acetate — Infusion for volume expansion in the ICU
  Other Names: Ringerfundin / Sterofundin
  Arms: Ringer acetate

SUMMARY:
* By tradition hydroxyethyl starch (HES) is used to obtain fast circulatory stabilisation in critically ill.
* High molecular weight HES may, however, cause acute kidney failure in patients with severe sepsis.
* Now the low molecular weight HES 130/0.4 is the preferred colloid in Scandinavian intensive care units (ICU) and 1st choice fluid for patients with severe sepsis.
* HES 130/0.4 is largely unstudied in ICU patients.
* This investigator-initiated Scandinavian multicentre trial will be conducted to assess the effects of HES 130/0.4 on mortality and endstage kidney failure in patients with severe sepsis.
* The trial will provide important data to all clinicians who resuscitate septic patients.

DETAILED DESCRIPTION:
Fluid is the mainstay treatment in sepsis resuscitation, but the effects of different crystalloid and colloid solutions on outcome remain unknown.

Previously, a high molecular weight hydroxyethyl starch, HES 200, was used, but this was found to cause acute kidney failure in patients with severe sepsis. As kidney failure is an independent risk factor for death in these patients, HES 200 is not used anymore. In stead a lower molecular weight starch, HES 130, has been developed. Presently, this is the preferred colloid in Scandinavian intensive care units (ICU), but the effects of HES 130 in ICU patients are currently unknown. The proposed Scandinavian multicentre study will be conducted to assess if HES 130 contributes to acute kidney failure in patients with severe sepsis. As HES 130 is widely used, the trial will provide important safety data to clinicians who resuscitate septic patients.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who

* Undergo resuscitation in the ICU
* AND fulfillment within the previous 24 hours of the criteria for severe sepsis (SCCM/ACCP)
* AND consent is obtainable either from the patient or by proxy (physician and/or next of kin)

Exclusion Criteria:

The following patients will not be evaluated for inclusion:

* Age < 18 years old
* Previously randomised in the 6S trial
* Allergy towards hydroxyethyl starch or malic acid
* Treatment with > 1000 ml's of any synthetic colloid within the last 24 hours prior to randomisation
* Any form of renal replacement therapy
* Acute burn injury > 10% body surface area
* Severe hyperkalaemia, p-K > 6 mM
* Liver or kidney transplantation during current hospital admission
* Intracranial bleeding within current hospitalisation
* Enrollment into another ICU trial of drugs with potential action on circulation, renal function or coagulation
* Withdrawal of active therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mortality or dialysis-dependency | 90 days

SECONDARY OUTCOMES:
Mortality | 28 days
Mortality | 6 months
Mortality | 1 year
Severity organ failure assessment score | Day 5
  Excluding Glascow coma score
Days free of ventilation | 90 days
  Among survivors
Days free of dialysis | 90 days
  Among survivors
Serious adverse reactions | Followed up until ICU discharge; consequently the time frame will vary among patients
  Severe bleeding or severe allergic reactions
Need of dialysis/haemofiltration | Within 90 days
Need of ventilation | Within 90 days
Kidney failure | Followed up until ICU discharge; consequently the time frame will vary among patients
  Severity organ failure assessment score > 2 in the renal component
Hospital length of stay | 90 days
Coagulation analyses | 5 days
  At selected hospitals whole-blood and biochemical coagulation analyses constitute additional secondary endpoints
NGAL | 5 days
  At selected trial sites will plasma and urinary NGAL be analysed at randomisation to assess the predictive value for dialyse and kidney failure

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD, PhD, Principal Investigator — ICU, Rigshospitalet, University of Copenhagen; Nicolai Haase, MD, Study Director — Rigshospitalet, Denmark
Locations (26):
- Denmark (18):
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hosptial, Copenhagen
  - Glostrup Hospital, Copenhagen
  - Herlev Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Herning Hospital, Herning
  - Hillerød Hospital, Hillerød
  - Hjørring Hospital, Hjørring
  - Holbæk Hospital, Holbæk
  - Holstebro Hospital, Holstebro
  - Køge Hospital, Køge
  - Næstved Hospital, Næstved
  - Odense University Hospital, Odense
  - Slagelse Hospital, Slagelse
  - Sønderborg Hospital, Sønderborg
  - Vejle Hospital, Vejle
- Finland (3):
  - Dept of Intensive Care, Helsinki University Hospital, Helsinki
  - Dept. of Intensive Care, Kuopio University Hospital, Kuopio
  - Dept of Intensive Care, Tampere University Hospital, Tampere
- Dept. of Intensive Care, Landspitali, Reykjavik, Iceland
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger
  - Intensive Care Unit, University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim University Hospital, Trondheim

REFERENCES:
- [Background] Perner A, Haase N, Wetterslev J, Aneman A, Tenhunen J, Guttormsen AB, Klemenzson G, Pott F, Bodker KD, Badstolokken PM, Bendtsen A, Soe-Jensen P, Tousi H, Bestle M, Pawlowicz M, Winding R, Bulow HH, Kancir C, Steensen M, Nielsen J, Fogh B, Madsen KR, Larsen NH, Carlsson M, Wiis J, Petersen JA, Iversen S, Schoidt O, Leivdal S, Berezowicz P, Pettila V, Ruokonen E, Klepstad P, Karlsson S, Kaukonen M, Rutanen J, Karason S, Kjaeldgaard AL, Holst LB, Wernerman J; Scandinavian Critical Care Trials Group. Comparing the effect of hydroxyethyl starch 130/0.4 with balanced crystalloid solution on mortality and kidney failure in patients with severe sepsis (6S--Scandinavian Starch for Severe Sepsis/Septic Shock trial): study protocol, design and rationale for a double-blinded, randomised clinical trial. Trials. 2011 Jan 27;12:24. doi: 10.1186/1745-6215-12-24. PMID 21269526
- [Result] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Derived] Ostrowski SR, Haase N, Muller RB, Moller MH, Pott FC, Perner A, Johansson PI. Association between biomarkers of endothelial injury and hypocoagulability in patients with severe sepsis: a prospective study. Crit Care. 2015 Apr 24;19(1):191. doi: 10.1186/s13054-015-0918-5. PMID 25907781
- [Derived] Perner A, Haase N, Winkel P, Guttormsen AB, Tenhunen J, Klemenzson G, Muller RG, Aneman A, Wetterslev J. Long-term outcomes in patients with severe sepsis randomised to resuscitation with hydroxyethyl starch 130/0.42 or Ringer's acetate. Intensive Care Med. 2014 Jul;40(7):927-34. doi: 10.1007/s00134-014-3311-y. Epub 2014 May 8. PMID 24807084
- [Derived] Muller RG, Haase N, Wetterslev J, Perner A. Effects of hydroxyethyl starch in subgroups of patients with severe sepsis: exploratory post-hoc analyses of a randomised trial. Intensive Care Med. 2013 Nov;39(11):1963-71. doi: 10.1007/s00134-013-3090-x. Epub 2013 Sep 14. PMID 24037226
- See also: Statistical analysis plan for the 6S trial — http://ssai.info/news/6s-trial-analysis-plan.html